CLINICAL TRIAL: NCT03598829
Title: A Prospective Clinical Trial Comparing Serum Mast Cell Tryptase (SMCT) Levels to Arthrofibrosis Rates Among Primary Total Knee Arthroplasty (TKA) Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 18-004103
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis; Arthropathy of Knee; Arthrofibrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Total Knee Arthroplasty: All patients enrolled in this study were part of the same recruitment group who whose SMCT levels will be observed pre and postoperatively. Primary TKA patients are having their native knee replaced.
  Interventions: Diagnostic Test: Tryptase, Serum test

INTERVENTIONS:
Diagnostic Test: Tryptase, Serum test — Blood draw lab test which measures concentration of Tryptase in the sample. Tryptase is the one of the primary secretions of active mast cells and is used as a measure of inflammatory activity. Normal Reference Value: <11.5 ng/mL
  Other Names: Serum Tryptase; Tryptase, S; TRYPT; Mast Cell Tryptase; CPT Code 83520

SUMMARY:
This research is being done to see if the amount of an enzyme in blood (called serum mast cell tryptase) changes before and after surgery. The investigators would like to see if these amounts are related to knee stiffness and pain in subjects that undergo a total knee replacement.

DETAILED DESCRIPTION:
Arthrofibrosis (AF), characterized by pain and limited mobility, affects a notable percentage of patients post-total knee arthroplasty (TKA). Despite various treatment advancements, the condition remains challenging to manage. Prior research has indicated a relationship between elevated serum mast cell tryptase (SMCT) levels and increased fibrosis in animal models, suggesting that SMCT could serve as a biomarker for arthrofibrosis in humans. This study aims to 1) assess pre- and postoperative SMCT levels in TKA patients, 2) evaluate SMCT's association with arthrofibrosis and clinical outcomes, and 3) determine the impact of allergic or inflammatory co-morbidities on SMCT levels.

ELIGIBILITY:
Inclusion Criteria:

* Investigators will include all patients with osteoarthritis who are surgical candidates for primary TKA. Investigators will include all eligible male or female patients between the ages of 20 years to 100 years old. All included study participants must be able to give an informed consent.

Exclusion Criteria:

* Significant femoral or tibial deformity due to congenital or traumatic etiologies, inflammatory arthritis, post-septic arthritis, osteomyelitis, prior infection of knee joint, osteoporosis, dislocated or fragmented patella
* Patients taking mast cell inhibitors and/or degranulation inhibitors for any reason.
* The presence of infections, highly communicable diseases (e.g. AIDS), active tuberculosis, venereal disease, hepatitis.
* Significant neurological or musculoskeletal disorders or disease that may adversely affect normal gait or weight bearing.
* Presence of previous prosthetic knee replacement devices (of any type)
* Metastatic disease
* Psychiatric illness
* Drug or alcohol abuse
* Inability to participate in standard postoperative rehabilitation protocol

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females between the ages of 20 to 100 years who are surgical candidates for primary total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Serum mast cell tryptase values | 1 year
  Serum mast tryptase values will be assessed pre and postoperatively to evaluate changes that can be expected in patients who are undergoing total knee replacement.
Evaluate serum mast cell tryptase association with arthrofibrosis | 1 year
  For patients who developed arthrofibrosis after total knee replacement, we will examine if a significant change in serum mast cell tryptase accompanies this outcome. This will help evaluate if tryptase levels may be useful as a marker of risk for arthrofibrosis.

SECONDARY OUTCOMES:
Evaluate the impact of allergic or inflammatory co-morbidities on serum mast cell tryptase levels | 1 year
  We will aim to examine to what extent allergic or inflammatory conditions influence changes in serum mast cell tryptase levels for patients undergoing total knee replacement. This aids in determining if underlying patient health affects how useful tryptase measurements could be as a marker for risk of arthrofibrosis, or if there is an association between these conditions and increased risk for arthrofibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abdel, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, as Mayo Clinic is the only institution involved in this research study and results reporting will be done via summary metrics and statistical analysis. Research participants did not consent for IPD to be shared outside of Mayo Clinic.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials